CLINICAL TRIAL: NCT00000804
Title: A Randomized Trial of L-735,524, An Inhibitor of the HIV Protease Enzyme, and Interleukin-2 in Persons Infected With HIV (NOTE: Only For Patients Who Previously Completed NIAID 93 CC-113)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: L DRUG
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2003-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Indinavir

INTERVENTIONS:
Drug: Indinavir sulfate

SUMMARY:
The purpose of this trial is to study L-735,524, which is an inhibitor of the HIV protease enzyme. It will be used with interleukin-2 in patients infected with HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)